CLINICAL TRIAL: NCT04018274
Title: A PHASE 1, RANDOMIZED, OPEN LABEL, 2 WAY CROSSOVER STUDY TO DEMONSTRATE A LACK OF AN EFFECT OF MULTIPLE DOSE PF 06651600 ON THE PHARMACOKINETICS OF SINGLE DOSE ORAL CONTRACEPTIVE STEROIDS IN HEALTHY FEMALE PARTICIPANTS
Brief Title: Effect of PF-06651600 on the Pharmacokinetics of Oral Contraceptive Steroids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7981035
Record Dates: First submitted 2019-07-11; First posted 2019-07-12 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Healthy
MeSH Terms: interventions — PF-06651600; Ethinyl Estradiol; Levonorgestrel; Contraceptives, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): In Treatment Sequence 1, period 1, participants will be dosed with a single administration of oral contraceptive (OC). Participants will continue directly into Period 2 where they will receive PF-06651600 PO for 9 days followed by administration of a single dose of OC on the morning of Day 10.
  Interventions: Drug: PF-06651600; Drug: Ethinyl estradiol (EE) and levonorgestrel(LN)
- Sequence 2 (Experimental): In Treatment Sequence 2, Period 1, participants will be dosed with PF-06651600 PO QD for 9 days and administered a single dose of OC on the morning of Day 10. After a washout period of at least 10 days, participants will continue into Period 2 and will receive an additional single dose of OC.
  Interventions: Drug: PF-06651600; Drug: Ethinyl estradiol (EE) and levonorgestrel(LN)

INTERVENTIONS:
Drug: PF-06651600 — 50 mg by mouth (PO) once daily (QD)
Drug: Ethinyl estradiol (EE) and levonorgestrel(LN) — Oral tablet containing 30 ug EE and 150 ug of LN
  Other Names: Oral contraceptives

SUMMARY:
This is a Phase 1, randomized, 2 way crossover, open-label study of the effect of multiple-dose PF 06651600 on single-dose oral contraceptive (OC) pharmacokinetics (PK) in healthy female subjects. Subjects will be randomized to 1 of 2 treatment sequences. A total of 28 healthy female subjects (14 in each treatment sequence) will be enrolled in the study. Each treatment sequence will consist of 2 periods.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Age and Sex:

1. Female participants of non childbearing potential who, at the time of screening, are between the ages of 18 and 60 years, inclusive.
2. Female participants who are healthy as determined by medical evaluation including detailed medical history, full physical examination, including blood pressure (BP) and pulse rate measurement, 12 lead ECG, or clinical laboratory tests.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Body mass index (BMI) of 17.5 to 35 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy, appendectomy).
3. Known immunodeficiency disorder, including positive serology for human immunodeficiency virus (HIV) at screening, or a first-degree relative with a hereditary immunodeficiency.
4. Infection with hepatitis B or hepatitis C viruses -

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 29 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for EE | predose, 30 minutes and 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post OC dose in Periods 1 and 2
  30 micrograms administered as oral OC combination tablet
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for LN | predose, 30 minutes and 1, 1.5, 2, 4, 6, 8, 12, 24, 36, 48, 72 and 96 hours post OC dose in Periods 1 and 2
  150 micrograms administered as oral OC combination tablet

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Quotient Sciences Screening Office, Coral Gables, Florida
  - Quotient Sciences, Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981035